CLINICAL TRIAL: NCT01754558
Title: One Year Outcome Using the Ajust System for Treatment of Urinary Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Martin Rudnicki, Ass. Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-252
Record Dates: First submitted 2011-12-28; First posted 2012-12-21 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (2):
- Ajust sling (Experimental): The sling a a new device for stress urinary incontinence. The sling is ajustable and is not penetrating the skin, i.e. is only attached to the obturator membrane
  Interventions: Procedure: Ajust system; Procedure: TVT/TVT-O
- TVT/TVT-O, polypropylne slings (Experimental): TVT/TVT-O system. These two systems is wellknown and used for treatment of stress urinary incontinence. The sling penetrate the skin in order to secure adjustment.
  Interventions: Procedure: Ajust system; Procedure: TVT/TVT-O

INTERVENTIONS:
Procedure: Ajust system — The use of Ajust system for stress incontinence
Procedure: TVT/TVT-O — sling surgery

SUMMARY:
During the last decade numerous new procedures have been presented regarding surgical treatment of urinary stress incontinence (1,2). Development of the midurethral tape procedure (TVT) changed the surgical procedure dramatically both regarding the extent of the surgical procedure and also decreased the morbidity remarkably. The success rate of the TVT procedure has been proven to be high (1,2 ). However, the development of the TOT/TVT-O procedures disclosed a new fixation point and further decreased the risk of bladder injury (1,2). Since the introduction of trans-obturator slings several mini-slings have been introduced in order to reduce the need of perforation of the skin and muscles (3,4,5). Although some systems seem promising (5) others have disclosed a long learning curve, pain problems following the procedure and lower success rates, compared to the traditional sling procedures. None of these mini-slings have been adjustable.

Recently the Ajust system for treatment of stress urinary incontinence was introduced. The system is a single incision sling procedure and consists of an adjustable Polypropylene mesh sling with self fixation anchors (6). In a feasibility study (6), the 6 months objective cure rate was 82%, but there is a lack of information regarding adverse events and durability of treatment success. Our preliminary experiences suggest, that the procedure has a rapid learning curve, low pain scores postoperatively and a 94% cure rate at 3 months follow-up (personal observation). Recently, several abstracts have indicated that the cure rate obtained by Ajust is comparable to TVT or TVT-O (10-12).

The purpose of the present study is (primary outcome):

To test the hypothesis that the Ajust and TVT, TVT-O and TOT, respectively are equal regarding subjective cure rate (cure is defined as subjectively not incontinent at all), i.e. the study is designed as a non-inferiority study. The study is performed as a randomised controlled trial without blinding. The study is powered to detect a 9% difference between the two groups. The subjective cure rate is based on ICIQ measurement

Secondary outcome:

* To test the hypothesis that Ajust is associated with a significantly lower postoperative pain perception.
* To test the hypothesis that antibiotic treatment is not necessary

DETAILED DESCRIPTION:
Primary endpoint: A cured patients is defined as no subjective symptoms (ICIQ-UI SF and ICIQ-OAB) and no objective detectable urinary leakage during coughing (300cc in the bladder and no leakage during coughing)

Secondary outcome: Pain-perception is evaluated by VAS scoring daily during the first postoperative week, including assessing the need for painkilling medication

The endpoint regarding the use of antibiotics is based on the number of urinary tract infections and infections related to the vaginal closure during the first postoperative months. All patients will evaluated postoperative by physical examination and by urinary dipstick

ELIGIBILITY:
Inclusion Criteria:

- 1. A medical history of stress urinary incontinence, i.e. leakage during coughing, sneezing or leakage during physical exertion. OR 2. A medical history of mixed urinary stress incontinence defined as complaint of involuntary leakage associated with urgency and stress incontinence. Stress incontinence has to the dominating symptom defined as more episodes of leakage due to coughing or physical exertion than with urgency.

3. A provocative stress test up to ten coughs at a standardized bladder volume (300 ml) confirming urinary leakage from the urethra while the patient is asked to cough or perform a Valsalva manoeuvre standing or lying (7). Furthermore, the patient has to present hypermobility of the urethra/bladder neck defined as significant downward rotation when coughing or during Valsalva.?

Exclusion Criteria:

1. Previous anti-incontinence surgery.
2. Residual urine volume >100 ml
3. Bladder capacity <200ml according to diary.
4. Planned or current pregnancy
5. Repeated urinary tract infections (>4 cystitis last year )
6. Current anticoagulation therapy that can´t be interrupted in due time prior to surgery
7. Known abnormal coagulation
8. Allergy to local anaesthetics
9. Co-existing pelvic pathology, such as ovarian mass etc
10. Vaginal POPQ anterior prolapse grade >=2
11. A medical history of predominantly urge urinary incontinence.
12. Patients unable to understand the protocol and a follow up
13. Patients younger than 18 and above or equal to 60 years.
14. Known or suspected neurological condition
15. Patients who have not paused acethylsalicylic acid (ASA) medication 7 days prior to surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
A change in number of cured patients | Up to 1 year
  Primary endpoint: A change in number of cured patients. The number of patients cured is anticipated to be equal in each group.
  A cured patients is defined as having no subjective symptoms (i.e. no scores on the ICIQ-UI SF and ICIQ-OAB) and no objective detectable urinary leakage during coughing (300cc in the bladder and no leakage during coughing.

SECONDARY OUTCOMES:
Pain-perception following surgery | Evaluated the first week following surgery, and at three and 12 months follow-up
  Secondary outcome: Pain-perception is evaluated by VAS scoring daily during the first postoperative week, including assessing the need for painkilling medication
  The endpoint regarding the use of antibiotics is based on the number of urinary tract infections and infections related to the vaginal closure during the first postoperative months. All patients will evaluated postoperative by physical examination and by urinary dipstick

OTHER OUTCOMES:
number of urinary tract infections and infections related to the vaginal closure during the first postoperative months. | Evaluated during the first week of follow-up and at 3 months follow-up
  The endpoint regarding the use of antibiotics is based on the number of urinary tract infections and infections related to the vaginal closure during the first postoperative months. All patients will evaluated postoperative by physical examination and by urinary dipstick

CONTACTS AND LOCATIONS:
Locations (1):
- Martin Rudnicki, Roskilde, Roskilde, Denmark

REFERENCES:
- [Derived] Temtanakitpaisan T, Buppasiri P, Lumbiganon P, Laopaiboon M, Rattanakanokchai S. Prophylactic antibiotics for preventing infection after continence surgery in women with stress urinary incontinence. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD012457. doi: 10.1002/14651858.CD012457.pub2. PMID 35349162
- [Derived] Rudnicki M, von Bothmer-Ostling K, Holstad A, Magnusson C, Majida M, Merkel C, Prien J, Jakobsson U, Teleman P. Adjustable mini-sling compared with conventional mid-urethral slings in women with urinary incontinence. A randomized controlled trial. Acta Obstet Gynecol Scand. 2017 Nov;96(11):1347-1356. doi: 10.1111/aogs.13205. Epub 2017 Sep 15. PMID 28815547